CLINICAL TRIAL: NCT04730141
Title: Effect of Mobilization Protocol on Mobilization Start Time and Patient Care Results in Patients Undergoing Abdominal Surgery
Brief Title: Effect of Mobilization Protocol on Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Fadime Koyuncu, Research Assistant, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 19208
Record Dates: First submitted 2021-01-22; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Abdominal Surgery; Nursing
Keywords: surgery and mobilization; early mobilization protocol

STUDY DESIGN:
Intervention Model Description: quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobilization protocol (Experimental): The early mobilization protocol developed by using up-to-date guidelines and expert opinions were applied to the patients in the intervention group.
  Interventions: Other: Patient mobilization with pre-operative mobilization training and mobilization protocol
- routine care (No Intervention): The routine mobilization follow-up approach of the intensive care unit was applied to the patients in the control group .

INTERVENTIONS:
Other: Patient mobilization with pre-operative mobilization training and mobilization protocol — Postoperative mobilization for the first 24 hours
  Arms: mobilization protocol

SUMMARY:
The aim of this study is to determine the effect of early mobilization protocol on patients' mobilization status and patient care outcomes in patients who undergo major abdominal surgery. This study is a prospective non-randomized controlled clinical trial.

DETAILED DESCRIPTION:
The study sample consisted of 42 patients, 21 of whom were the control group and 21 were the intervention group, who had undergone major abdominal open surgery between May and September 2019. The routine mobilization follow-up approach of the intensive care unit was applied to the patients in the control group, and the early mobilization protocol developed by using up-to-date guidelines and expert opinions were applied to the patients in the intervention group. In the study, the data of the control group were firstly collected, then the early mobilization protocol was introduced to the patients through the training brochure prepared and then data of the intervention group were collected. In the study, the characteristics of the patients in both groups belonging to the preoperative period, the distance they walked in the 6-minute walking test and the results of the postoperative period were recorded.

ELIGIBILITY:
Inclusion Criteria:

* To undergo major abdominal open surgery
* ASA <IV
* Being over the age of 18
* Not having a barrier to communication
* Having agreed to participate in the study

Exclusion Criteria:

* Being diagnosed that may limit mobilization
* Being diagnosed with chronic obstructive pulmonary disease
* ASA IV-V-VI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
The effect of mobilization protocol on mobilization start time | first 24 hours postoperatif
  In the postoperative period, the hour of mobilization of the patient was recorded.The group in which the mobilization protocol was applied and the group in which the mobilization protocol was not applied were compared
Postoperative sleep quality | Postoperative 24th hour
  VAS is considered a valid, reliable and usable measurement tool used to convert some values that cannot be measured numerically into numericals. Possible scores from 0 (worst case) to 10 (best case)
Postoperative patient satisfaction | Postoperative 24th hour
  VAS is considered a valid, reliable and usable measurement tool used to convert some values that cannot be measured numerically into numericals. Possible scores from 0 (worst case) to 10 (best case)

SECONDARY OUTCOMES:
Postoperative number of steps | The total number of steps taken during the first 24 hours postoperatively
  Pedometer programs are easy-to-use mobile applications where features such as the number of steps taken at a given time and walking distance can be recorded. Pedometer application is downloaded to the phone, the number of steps and walking distance are recorded by carrying it in a pocket or bag. In this study, Developer: ITO Technologies Inc, category: health and fitness, version 1.1.10 pedometer program was used.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Iyiun, Study Director — Gulhane Hemsirelik Fakultesi
Locations (1):
- Fadime, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No